CLINICAL TRIAL: NCT00413335
Title: Effects of Rosiglitazone on the Metabolic Phenotype of Impaired Glucose Tolerance in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Sonia Caprio, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0508000532
Record Dates: First submitted 2006-12-15; First posted 2006-12-19 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Obesity; Impaired Glucose Tolerance; Type 2 Diabetes Mellitus
Keywords: Childhood and Adolescent Obesity; Metabolic phenotype; Impaired Glucose Tolerance; Type 2 Diabetes Mellitus; Insulin Sensitivity; Insulin Resistance; Abdominal fat partitioning; Impaired Glucose Tolerance (IGT); Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Obesity; Glucose Intolerance; Diabetes Mellitus, Type 2; Pediatric Obesity; Insulin Resistance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subject undergoes ogtt, hyperinsulinemic-euglycemic clamp, abdominal and liver MRI, NMR and DEXA scan. Subject then receives Rosiglitazone. Subjects are followed every 2 weeks. Imaging repeated at 2 months. 12 week follow up. And then all tests are repeated at 4 months.
  Interventions: Drug: Rosiglitazone
- 2 (Placebo Comparator): Subject has ogtt, hyperinsulinemic-euglycemic clamp, abdominal and liver MRI, DEXA, NMR. Subject is randomized (double-blind) to placebo. Is followed every 2 weeks, repeats imaging at 2 months, is seen at 12 weeks and then repeats all tests at 2 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone — 2mg to begin then 4mg, twice daily for 4 months
  Other Names: Avandia
  Arms: 1
Drug: Placebo — Subject receives placebo.
  Arms: 2

SUMMARY:
The purpose of the study is to determine whether treatment of children and adolescents with Impaired Glucose Tolerance (IGT) with rosiglitazone will lead to improvements in insulin sensitivity and glucose tolerance.

DETAILED DESCRIPTION:
Impaired Glucose Tolerance (IGT) is a prelude to diabetes, which is increasing in prevalence in obese children and adolescents with marked obesity. This condition tends to progress to Type 2 Diabetes Mellitus (T2DM) at an alarmingly rapid tempo. The increased prevalence of childhood and adolescent obesity and greater risk of IGT, and progression to diabetes, in this population set the stage for a series of studies aimed at understanding the metabolic phenotype and natural history of pre-diabetes in obese youth. The investigators found that obese children and adolescents with IGT are characterized by marked insulin resistance related to altered lipid partitioning, favoring lipid deposition in the visceral and intramyocellular compartment. Furthermore, the investigators found an impairment of the acute insulin response in these youngsters. Follow-up revealed a rapid deterioration from IGT to frank diabetes. Based on these studies, there is a strong rationale for changing the balance between visceral and subcutaneous fat and muscle lipid content in a more favorable pattern in order to improve insulin sensitivity.

The primary objective of this study is to determine, in a group of ethnically diverse children and adolescents with IGT, whether treatment with rosiglitazone leads to improvements in insulin sensitivity and glucose tolerance. Secondary objectives are to determine whether rosiglitazone is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Aged 10 to 18 yrs (females: Tanner stage II-V;and males:testes size>6ml)
* IGT based on 2-hr plasma glucose>140mg/dl and <200mg/dl during an OGTT.

Exclusion Criteria:

* Baseline creatinine>1.0mg
* AST and ALT>2.5 ULN
* Anemia (Hct<30)
* Pregnancy (females must have a negative urine pregnancy test during the study)
* Cardiac or pulmonary or other significant chronic illness
* Plans to increase the frequency or intensity of a regular exercise program
* Psychiatric disorder or substance abuse of anorexic agents.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Caprio, MD, Principal Investigator — Yale School of Medicine Department of Pediatric Endocrinology
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a multi-ethnic cohort of obese children and adolescents drawn from the Pediatric Obesity Clinic at Yale-New Haven Hospital.
Pre-assignment Details: Obese children and adolescents with positive risk factors for Type 2 Diabetes (T2DM) were screened by using a standard oral glucose tolerance test (OCTT).
Groups:
- Active Arm (Rosiglitazone): Subject undergoes ogtt, hyperinsulinemic-euglycemic clamp, abdominal and liver MRI, NMR and DEXA scan. Subject then receives Rosiglitazone. Subjects are followed every 2 weeks. Imaging repeated at 2 months. 12 week follow up. And then all tests are repeated at 4 months.
  Rosiglitazone : 2mg to begin then 4mg, twice daily for 4 months
- Inactive Arm (Placebo): Subject has ogtt, hyperinsulinemic-euglycemic clamp, abdominal and liver MRI, DEXA, NMR. Subject is randomized (double-blind) to placebo. Is followed every 2 weeks, repeats imaging at 2 months, is seen at 12 weeks and then repeats all tests at 2 months.
  Placebo : Subject receives placebo.
Period: Overall Study
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo)
Started | 12 | 9
Completed | 12 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo) | Total
Number analyzed (Participants) | 12 | 9 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 12.8 (1.6) | 13.9 (2.0) | 13.0 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in Whole-body Insulin Sensitivity
Description: This describes the percent changes in insulin sensitivity. Insulin sensitivity was expressed as whole body insulin sensitivity index (WBISI) which is based on the values of insulin (microunits per milliliter) and glucose (milligrams per deciliter) obtained from the OGTT and the corresponding fasting values.The formula is: WBISI=10.000/square root of (fasting glucose x fasting insulin)x(mean glucose x mean insulin).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo)
Number analyzed (Participants) | 12 | 9
percentage of change from baseline | 87.4 (77.0) | 63.1 (61.6)

2. Primary Outcome: Mean Percent Change in Visceral-to-subcutaneous Abdominal Fat
Description: This describes the percent changes of the ratio between visceral and subcutaneous abdominal fat.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo)
Number analyzed (Participants) | 12 | 9
percentage of change from baseline | -7.3 (23.1) | 8.9 (22.6)

3. Primary Outcome: Percentage of Subjects Who Converted Impaired Glucose Tolerance (IGT) to Normal Glucose Tolerance (NGT)
Description: This refers to the number of subjects that converted from IGT to NGT. NGT is defined as fasting glucose lower than 100 mg/dl and 2 hours glucose lower than 140 mg/dl. IGT is defined as 2 hours glucose higher than 140 mg/dl.
Time Frame: 4 months
Measure: Number; unit: percentage of participants
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo)
Number analyzed (Participants) | 12 | 9
percentage of participants | 58 | 44

4. Secondary Outcome: Mean Percent Change From Baseline in Adiponectin
Description: This refers to the changes of adiponectin levels.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo)
Number analyzed (Participants) | 12 | 9
percentage of change from baseline | 79.3 (78.2) | 19.8 (52.8)

5. Primary Outcome: Mean Percent Change From Baseline in Hepatic Fat Fraction (HFF)
Description: It refers to the percent changes of hepatic fat content.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo)
Number analyzed (Participants) | 12 | 9
percentage of change from baseline | 2.7 (107) | 81 (267)

ADVERSE EVENTS:
Arm/Group | Active Arm (Rosiglitazone) | Inactive Arm (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes